CLINICAL TRIAL: NCT01923090
Title: An Open Label Study of 5α-reductase Inhibition on the Regulation of Insulin Action and Metabolic Phenotype in Healthy Volunteers.
Brief Title: Finasteride, Dutasteride and Insulin Action
Acronym: FIND-IT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Principal Investigator, Dr Jeremy Tomlinson, MRC Senior clinical fellow and Reader in Endocrinology, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_12-098; 12/WM/0122 (Other: South Birmingham Local Research Ethics committee)
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Finasteride; Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Finasteride (Experimental): Finasteride treatment 5mg for 3 weeks
  Interventions: Drug: Finasteride
- Dutasteride (Experimental): Dutasteride treatment 0.5mg for 3 weeks
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Finasteride — Finasteride 5mg once daily for 3 weeks
  Arms: Finasteride
Drug: Dutasteride — Dutasteride 0.5mg once daily for 3 weeks
  Arms: Dutasteride

SUMMARY:
The purpose of this study is to see if an enzyme in the body (5-alpha reductase, 5αR) is important in controlling how the body handles sugar and fat. The investigators believe that 5αR is a crucial step in regulating these actions as well as controlling how insulin works in the body but regulating the amount of steroid hormones including cortisol and testosterone in the body. In previous clinical studies, the investigators have shown that the activity of 5αR increases as you gain weight and decreases with weight loss. In addition, work that the investigators have performed in the laboratory has shown that if you increase 5αR levels in liver cell grown in the laboratory, the amount of fat that they contain increases. The investigators would therefore like to demonstrate the effect of inhibition 5αR on the regulation of insulin, glucose and fat in the body.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18-65years
* BMI 20-35kg/m2
* BMI >35kg/m2

Exclusion Criteria:

* Diabetes Mellitus
* Glucocorticoid use within the last 6 months
* Uncontrolled hypertension (BP>160/100mmHg)
* Drugs know to impact upon glucocorticoid metabolism

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity | 3 weeks
  stable isotope measurements of glucose production rate and glucose disposal

SECONDARY OUTCOMES:
adipose tissue insulin sensitivity | 3 weeks
  insulin mediated suppression of glycerol release into adipose tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Wellcome Trust Clinical Research Facility, Queen Elizabeth Hospital, Birmingham, West Midlands, United Kingdom